CLINICAL TRIAL: NCT01641692
Title: A Multi-national, Randomized, Double-blind, Placebo-controlled, 3-period Crossover Study With GSK 573719 as Monotherapy in Adult Subjects With Asthma
Brief Title: A 3-period Crossover Study With GSK573719 as Monotherapy in Adult Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 116402
Record Dates: First submitted 2012-05-31; First posted 2012-07-17 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Asthma
Keywords: Asthma; Pharmacokinetics; GSK573719; Adults; Pharmacogenetics
MeSH Terms: conditions — Asthma | interventions — GSK573719; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- GSK573719 15.6 mcg (Experimental): GSK573719 (Umeclinidium bromide) 15.6 mcg once-daily
  Interventions: Drug: GSK573719 Active treatment or Placebo; Procedure: GSK573719 (Sub-group cohort); Drug: Salbutamol/Albuterol
- GSK573719 31.25 mcg (Experimental): GSK573719 (Umeclinidium bromide) 31.25 mcg once-daily
  Interventions: Drug: GSK573719 Active treatment or Placebo; Procedure: GSK573719 (Sub-group cohort); Drug: Salbutamol/Albuterol
- GSK573719 62.5 mcg (Experimental): GSK573719 (Umeclinidium bromide) 62.5 mcg once-daily
  Interventions: Drug: GSK573719 Active treatment or Placebo; Procedure: GSK573719 (Sub-group cohort); Drug: Salbutamol/Albuterol
- GSK573719 125 mcg (Experimental): GSK573719 (Umeclinidium bromide) 125 mcg once-daily
  Interventions: Drug: GSK573719 Active treatment or Placebo; Procedure: GSK573719 (Sub-group cohort); Drug: Salbutamol/Albuterol
- GSK573719 250 mcg (Experimental): GSK573719 (Umeclinidium bromide) 250 mcg once-daily
  Interventions: Drug: GSK573719 Active treatment or Placebo; Procedure: GSK573719 (Sub-group cohort); Drug: Salbutamol/Albuterol
- GSK573719 15.6 mcg twice-daily (Experimental): GSK573719 (Umeclinidium bromide) 15.6 mcg twice-daily
  Interventions: Drug: GSK573719 Active treatment or Placebo; Procedure: GSK573719 (Sub-group cohort); Drug: Salbutamol/Albuterol
- GSK573719 31.25 mcg twice daily (Experimental): Gsk573719 (Umeclinidium bromide) 31.25 mcg twice-daily
  Interventions: Drug: GSK573719 Active treatment or Placebo; Procedure: GSK573719 (Sub-group cohort); Drug: Salbutamol/Albuterol
- Matched Placebo (Placebo Comparator): Matched Placebo arm
  Interventions: Drug: GSK573719 Active treatment or Placebo; Procedure: GSK573719 (Sub-group cohort); Drug: Salbutamol/Albuterol

INTERVENTIONS:
Drug: GSK573719 Active treatment or Placebo — Eligible subjects will be randomised to a sequence of three treatments from 8 possible arms: 7 active drug doses (15.6mcg, 31.25 mc, 62.5mcg 125mcg or 250mcg GSK573719 once daily; 15.6mcg or 31.25 mcg GSK573719 taken twice daily) or matched placebo.
Procedure: GSK573719 (Sub-group cohort) — Subjects at selected Sub-group sites (approximately 30% of the total population) will have additional serial assessments and procedures (including blood and urine samples for pharmacokinetic analysis) at the start (Day 1) and at the end (Days 14 and 15) of each treatment period. On Day 14 of each treatment period subjects will remain overnight at the clinic for 24-hour assessments, including spirometry, ECGs, and 24-hour Holter monitoring.
Drug: Salbutamol/Albuterol — Salbutamol/Albuterol, short-activing beta agonist provided to all subjects to be taken as needed for the relief of asthma symptoms.throughout the study period, including washout periods

SUMMARY:
This is a multi-national, randomized, double-blind, 3-period crossover, incomplete block design to evaluate 5 once-daily and 2 twice-daily doses of GSK573719 in combination with placebo. The study will explore the dose range of GSK573719 in asthmatic subjects who are currently using non-ICS controller medications. Subjects will participate in the study for up to a maximum of 14 weeks. At randomization subjects will be stratified by age to ensure adequate exposure to GSK573719 throughout the expected age range. The primary endpoint will be trough FEV1 obtained 24 hours after the last morning dose on Day 14 of each treatment sequence.

A sub-group of subjects at selected sites (approximately 30% of the total population) will have additional serial assessments for spirometry, ECG and Holter, and pharmacokinetic sampling at the start and end of each treatment period. Safety assessments will include monitoring for adverse events, laboratory tests, asthma symptom assessments and twice daily PEF evaluation. Consenting subjects will have a blood sample taken for pharmacogenetic analysis.

DETAILED DESCRIPTION:
Asthma, a reversible obstructive disease of the airways, is defined as a chronic inflammatory disorder of the airways in which many of the cells and cellular mediators play a role. The chronic inflammation is associated with airway hyper-responsiveness that leads to recurrent episodes of wheezing, breathlessness, chest tightness, and coughing, particularly at night or early in the morning. These episodes are usually associated with widespread, but variable airflow obstruction within the lung that is often reversible either spontaneously or with treatment (NIH 2007, GINA, 2010,). Guidelines recommend a stepwise approach to the management of asthma. For many patients with mild disease, asthma symptoms can be adequately relieved by 'on demand' use of a short acting beta-2 -agonist (SABA) alone. A long-acting, inhaled, muscarinic receptor antagonist (LAMA) exerts its effects via distinct and complementary bronchodilator mechanisms on large and small airways through antagonism of the endogenous agonist acetylcholine at the muscarinic receptors leading to smooth muscle relaxation and bronchodilation. However, most experience with older anti-cholinergics has been with acute use and little is known about their effect in chronic use or as maintenance in asthma.

Newer more selective muscarinic receptor antagonists are being developed for chronic use which appear to have a better adverse event profile compared with older anti-cholinergics in the treatment of asthma [Moulton 2011]. A once daily long-acting, inhaled, muscarinic receptor antagonist (LAMA) bronchodilator, GSK573719, may offer an alternative treatment option to patients with asthma.

The proposed study is a multi-national, randomized, double-blind, 3-period crossover, incomplete block study in outpatient subjects with mild asthma and who are not using inhaled corticosteroids (ICS) for symptom control. The primary objective of this study is to evaluate the dose response, efficacy and safety of five once-daily doses of GSK573719 compared with placebo, over a 14-day treatment period, in patients with asthma. A placebo arm will be included to determine an absolute treatment effect over placebo for each GSK573719 dose regimen.

Each eligible subject will be randomized to receive 3 out of 8 potential treatments in sequence over a total of three 14-day treatment periods. There will be 12 clinic visits including a safety follow-up visit at the end of the study. All subjects will be provided with albuterol (salbutamol) for use on an 'as-needed' basis throughout the run-in, treatment and washout periods. A sub-group (approximately 30%) of the study population will comprise subjects from selected sites. These subjects will have additional assessments at the start and end of each treatment period, including serial spirometry, serial ECGs, 24 hour Holter monitoring, and samples of blood and urine for pharmacokinetic analysis. Other safety parameters include the incidence of adverse events, vital signs, clinical laboratory parameters, ECGs and spirometry, including twice daily peak expiratory flow, asthma exacerbation assessment. and use of salbutamol.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Outpatient (sub-group will have 3 overnight stays at clinic)
* Diagnosis of asthma (NIH 2007) for at least 6 months
* Male or Eligible female (females of child-bearing potential must use acceptable method of birth control)
* A best AM pre-bronchodilator FEV1 of 60% to 85% of predicted normal value at Screening
* Reversibility of disease demonstrated by at least 12% and 200mL increase in FEV1 .
* Subjects must have been prescribed a non-corticosteroid controller at least 3 months preceding Visit 1, and/or a short-acting beta 2 agonist, without the use of inhaled corticosteroids in the 4 weeks prior to Visit 1
* Subjects must be able to replace their current short-acting Beta-2-agonist with albuterol/salbutamol aerosol inhaler for the duration of the study
* Subjects must be judged capable of withholding albuterol/salbutamol for at least 4 hours prior to study visits

Exclusion Criteria:

* History of life threatening asthma
* Severe asthma exacerbation
* Respiratory infection within expected to affect subject's ability to participate
* Concurrent respiratory disease
* Current smoker or smoking history of 10 pack years or more
* Diseases preventing use of anticholinergics
* Other clinically significant, uncontrolled condition or disease which would pose a safety risk to the patient, or confound interpretation of study results
* Drug allergy to any Beta-2-agonist, sympathomimetic drug, intranasal, inhaled or systemic corticosteroid therapy
* Known or suspected sensitivity to the constituents of the Novel DPI (ie lactose)
* History of severe milk protein allergy
* Administration of prescription or over-the-counter medication that would significantly affect the course of asthma, or interact with the study drug
* Any infirmity, disability or disease of a child or family member likely to impair compliance
* Alcohol or substance abuse history
* Viral hepatitis B surface antigen or Hepatitis C antibody
* Known HIV-positive history.
* Affiliation with investigator or site staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (36):
- United States (12):
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, San Antonio, Texas
- Bulgaria (7):
  - GSK Investigational Site, Lovech
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Varna
- Germany (6):
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Mexico (2):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
- Peru (4):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, San Borja, Lima region
  - GSK Investigational Site, San Miguel, Lima region
  - GSK Investigational Site, Santiago de Surco, Lima region
- Poland (5):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Ruda Śląska
  - GSK Investigational Site, Zawadzkie
  - GSK Investigational Site, Zgierz

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lee LA, Briggs A, Edwards LD, Yang S, Pascoe S. A randomized, three-period crossover study of umeclidinium as monotherapy in adult patients with asthma. Respir Med. 2015 Jan;109(1):63-73. doi: 10.1016/j.rmed.2014.10.009. Epub 2014 Oct 28. PMID 25464907
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 116402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116402 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive a sequence of 3 of 8 possible treatments over 3 treatment periods. There are 56 combinations of 3 treatments from the 8 study treatments, each of which can be ordered in 6 ways (totaling 336 possible sequences; 246 were randomly assigned). Participant Flow data are presented by treatment rather than sequence.
Groups:
- Placebo: Participants received matching placebo in the morning via dry powder inhaler (DPI) A and in the evening via DPI B for 14 days.
- UMEC 15.6 µg QD: Participants received umeclidinium bromide (UMEC) 15.6 micrograms (µg) in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- UMEC 31.25 µg QD: Participants received UMEC 31.25 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- UMEC 62.5 µg QD: Participants received UMEC 62.5 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- UMEC 125 µg QD: Participants received UMEC 125 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- UMEC 250 µg QD: Participants received UMEC 250 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- UMEC 15.6 µg BID: Participants received UMEC 15.6 µg in the morning via DPI A and in the evening via DPI B for 14 days.
- UMEC 31.25 µg BID: Participants received UMEC 31.25 µg in the morning via DPI A and in the evening via DPI B for 14 days.
Period: Treatment Period 1
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Started | 42 | 45 | 51 | 41 | 43 | 39 | 38 | 51
Completed | 40 | 45 | 50 | 41 | 39 | 37 | 38 | 48
Not Completed | 2 | 0 | 1 | 0 | 4 | 2 | 0 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Protocol-defined Stopping Criteria | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Period: Washout Period 1 (12-14 Days)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Started | 40 | 45 | 50 | 41 | 39 | 37 | 38 | 48
Completed | 36 (Participants withdrawing during washout are counted under the last treatment taken.) | 44 (Participants withdrawing during washout are counted under the last treatment taken.) | 47 (Participants withdrawing during washout are counted under the last treatment taken.) | 39 (Participants withdrawing during washout are counted under the last treatment taken.) | 35 (Participants withdrawing during washout are counted under the last treatment taken.) | 37 (Participants withdrawing during washout are counted under the last treatment taken.) | 36 (Participants withdrawing during washout are counted under the last treatment taken.) | 47 (Participants withdrawing during washout are counted under the last treatment taken.)
Not Completed | 4 | 1 | 3 | 2 | 4 | 0 | 2 | 1
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol-defined Stopping Criteria | 1 | 0 | 3 | 1 | 3 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Started | 33 (By crossover design, participants were assigned to a different treatment arm in each period.) | 46 (By crossover design, participants were assigned to a different treatment arm in each period.) | 40 (By crossover design, participants were assigned to a different treatment arm in each period.) | 41 (By crossover design, participants were assigned to a different treatment arm in each period.) | 37 (By crossover design, participants were assigned to a different treatment arm in each period.) | 45 (By crossover design, participants were assigned to a different treatment arm in each period.) | 43 (By crossover design, participants were assigned to a different treatment arm in each period.) | 36 (By crossover design, participants were assigned to a different treatment arm in each period.)
Completed | 30 | 46 | 40 | 41 | 37 | 43 | 43 | 35
Not Completed | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol-defined Stopping Criteria | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Period: Washout Period 2 (12-14 Days)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Started | 30 | 46 | 40 | 41 | 37 | 43 | 43 | 35
Completed | 30 (Participants withdrawing during washout are counted under the last treatment taken.) | 46 (Participants withdrawing during washout are counted under the last treatment taken.) | 39 (Participants withdrawing during washout are counted under the last treatment taken.) | 41 (Participants withdrawing during washout are counted under the last treatment taken.) | 34 (Participants withdrawing during washout are counted under the last treatment taken.) | 42 (Participants withdrawing during washout are counted under the last treatment taken.) | 42 (Participants withdrawing during washout are counted under the last treatment taken.) | 34 (Participants withdrawing during washout are counted under the last treatment taken.)
Not Completed | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 1
Not completed — Protocol-defined Stopping Criteria | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Period: Treatment Period 3
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Started | 43 (By crossover design, participants were assigned to a different treatment arm in each period.) | 33 (By crossover design, participants were assigned to a different treatment arm in each period.) | 38 (By crossover design, participants were assigned to a different treatment arm in each period.) | 42 (By crossover design, participants were assigned to a different treatment arm in each period.) | 40 (By crossover design, participants were assigned to a different treatment arm in each period.) | 39 (By crossover design, participants were assigned to a different treatment arm in each period.) | 35 (By crossover design, participants were assigned to a different treatment arm in each period.) | 38 (By crossover design, participants were assigned to a different treatment arm in each period.)
Completed | 43 | 32 | 37 | 42 | 40 | 39 | 33 | 38
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol-defined Stopping Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3 or Follow-up
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Started | 43 | 32 | 37 | 42 | 40 | 39 | 33 | 38
Completed | 42 (Participants withdrawing during washout are counted under the last treatment taken.) | 32 (Participants withdrawing during washout are counted under the last treatment taken.) | 36 (Participants withdrawing during washout are counted under the last treatment taken.) | 41 (Participants withdrawing during washout are counted under the last treatment taken.) | 40 (Participants withdrawing during washout are counted under the last treatment taken.) | 37 (Participants withdrawing during washout are counted under the last treatment taken.) | 32 (Participants withdrawing during washout are counted under the last treatment taken.) | 38 (Participants withdrawing during washout are counted under the last treatment taken.)
Not Completed | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol-defined Stopping Criteria | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Treatments: The treatment phase was comprised of three 14-day treatment periods. Treatment Period 1 and 2 were followed by a 12-14 day washout period. Treatment Period 3 was followed by a 5 to 9 day washout period before the Follow-up visit. Participants were randomly assigned to receive a sequence of 3 of the 8 active treatments :
  UMEC 15.6, 31.25, 62.5, 125, 250 µg QD and UMEC 15.6, 31.25 µg BID, placebo.
Arm/Group | All Study Treatments
Number analyzed (Participants) | 350
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (14.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232
  Male | 118
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage (HER) | 33
  American Indian or Alaskan Native | 85
  Asian-Japanese/East Asian HER/South East Asian HER | 4
  White | 197
  American Indian or Alaskan Native & White | 31

OUTCOME MEASURES:

1. Primary Outcome: Final Dose-response Model for Trough Forced Expiratory Volume in One Second (FEV1)
Description: Dose-response was conducted for both QD and BID UMEC doses on trough FEV1 (measure of lung function, defined as the maximal amount of air that can be forcefully exhaled in 1 second) on D 15. Total daily dose of UMEC was used in the modeling. The null model was the final model. The null model is defined as: CFEV1,ij=(THETA1+ETA1j)*meanBL+(THETA2+ETA1j)*periodBL+EPSij, where CFEV1,ij represents the change from BL in trough FEV1 for participant j measured at period i. THETA1 and THETA2 were the slopes with respect to meanBL and periodBL, respectively. Omegas were the variance of the slopes on meanBL and periodBL (ETA1j, ETA2j) for each participant and Sigma was the variance of the residual errors (EPSij). MeanBL is the mean of the Baseline (BL) which is the FEV1 value recorded pre-dose on D 1 of each TP; periodBL is the difference between the BL and the meanBL in each TP for each participant.
Time Frame: Day 15 of each treatment period (up to Study Day 71)
Population: Intent-To-Treat (ITT) Population: : all participants randomized to treatment and who received at least one dose of study medication. All participants with >=1 post-Baseline assessment and non-missing covariate data are included in the analysis. The number of participants represents participants who provided data at Day 15.
Measure: Geometric Mean (95% Confidence Interval); unit: unitless
Arm/Group | All Study Treatments
Number analyzed (Participants) | 332
unitless
  Theta1 (mean Baseline) | 0.0363 [0.0280 to 0.0450]
  Theta2 (period Baseline) | -0.97 [-1.06 to -0.881]
  Omega (mean Baseline) | 0.00371 [0.002 to 0.005]
  Omega (period Baseline) | 0.149 [0 to 0.298]
  Sigma (Variance of Residual error) | 0.0393 [0.028 to 0.050]

2. Primary Outcome: Change From Baseline in Trough FEV1 on Day 15 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Treatment Day 15 is defined as the value obtained 24 hours after the morning dose administered on Day 14. Analysis was performed using a mixed model, including treatment, period, period Baseline FEV1 and mean Baseline FEV1 as fixed effects and participant as a random effect. Baseline is the FEV1 value recorded pre-dose on Day 1 of each treatment period; mean Baseline is the mean of the Baselines for each participant and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Change from Baseline for each treatment period is the trough FEV1 at Day 15 minus the Baseline value for that treatment period.
Time Frame: Day 15 of each treatment period (up to Study Day 71)
Population: ITT Population. All participants with >=1 post-Baseline assessment and non-missing covariate data are included in the analysis. The number of participants represents participants who provided data at Day 15.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Placebo: Participants received matching placebo in the morning via DPI A and in the evening via DPI B for 14 days.
- UMEC 15.6 µg QD: Participants received UMEC 15.6 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 110 | 120 | 124 | 122 | 113 | 117 | 113 | 118
Liters | 0.046 (0.0235) | 0.112 (0.0226) | 0.076 (0.0222) | 0.080 (0.0224) | 0.134 (0.0232) | 0.057 (0.0228) | 0.103 (0.0232) | 0.097 (0.0227)
Statistical Analysis 1: Comparison: Placebo vs UMEC 15.6 µg QD; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis; Mean Difference (Final Values) = 0.066, 95% CI 2-sided [0.004 to 0.127]
Statistical Analysis 2: Comparison: Placebo vs UMEC 31.25 µg QD; Test type: Superiority or Other; p = 0.331, Mixed Models Analysis; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [-0.030 to 0.090]
Statistical Analysis 3: Comparison: Placebo vs UMEC 62.5 µg QD; Test type: Superiority or Other; p = 0.272, Mixed Models Analysis; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [-0.027 to 0.095]
Statistical Analysis 4: Comparison: Placebo vs UMEC 125 µg QD; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = 0.088, 95% CI 2-sided [0.026 to 0.149]
Statistical Analysis 5: Comparison: Placebo vs UMEC 250 µg QD; Test type: Superiority or Other; p = 0.722, Mixed Models Analysis; Mean Difference (Final Values) = 0.011, 95% CI 2-sided [-0.050 to 0.073]
Statistical Analysis 6: Comparison: Placebo vs UMEC 15.6 µg BID; Test type: Superiority or Other; p = 0.076, Mixed Models Analysis; Mean Difference (Final Values) = 0.057, 95% CI 2-sided [-0.006 to 0.119]
Statistical Analysis 7: Comparison: Placebo vs UMEC 31.25 µg BID; Test type: Superiority or Other; p = 0.101, Mixed Models Analysis; Mean Difference (Final Values) = 0.051, 95% CI 2-sided [-0.010 to 0.113]

3. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Refer to the general Adverse AE/SAE module for a complete list of SAEs.
Time Frame: From Baseline until the end of Treatment Period 3 (up to Study Day 70)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
Participants
  Any AE | 15 | 12 | 13 | 21 | 26 | 28 | 16 | 12
  Any SAE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Participants With Asthma Exacerbations During the Treatment Period
Description: Worsening of asthma symptoms is monitored throughout the study. Severe exacerbation (deterioration of asthma requiring use of systemic corticosteroids for 3 days, inpatient hospitalization or emergency department visit due to asthma) is an exclusion criterion and requires withdrawal from the study. Asthma symptoms were assessed daily using an electronic diary throughout study.
Time Frame: From Baseline until the end of Treatment Period 3 (up to Study Day 70)
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
Participants | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1

5. Primary Outcome: Change From Baseline in Systolic Blood Pressure on Day 14 of Each Treatment Period
Description: Blood pressure measurement included systolic blood pressure (SBP). Blood pressure was measured in a sitting position after the participant was kept at rest for at least 5 minutes. Analysis was performed using a mixed model, including treatment, period, period Baseline and mean Baseline for the measure as fixed effects and participant as a random effect. Baseline is the value recorded pre-dose on Day 1 of each treatment period; mean Baseline is the mean of the Baselines for each participant and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Change from Baseline was calculated as the assessment value at Day 14 minus the Baseline value.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 112 | 122 | 127 | 123 | 114 | 119 | 114 | 122
Millimeters of mercury (mmHg) | -0.4 (0.71) | -0.6 (0.68) | -1.0 (0.67) | 1.1 (0.68) | -0.6 (0.71) | 0.0 (0.69) | 0.3 (0.71) | -1.2 (0.69)
Statistical Analysis 1: Comparison: Placebo vs UMEC 15.6 µg QD; Test type: Superiority or Other; p = 0.840, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.1 to 1.7]
Statistical Analysis 2: Comparison: Placebo vs UMEC 31.25 µg QD; Test type: Superiority or Other; p = 0.553, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.4 to 1.3]
Statistical Analysis 3: Comparison: Placebo vs UMEC 62.5 µg QD; Test type: Superiority or Other; p = 0.121, Mixed Models Analysis; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.4 to 3.3]
Statistical Analysis 4: Comparison: Placebo vs UMEC 125 µg QD; Test type: Superiority or Other; p = 0.814, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.1 to 1.7]
Statistical Analysis 5: Comparison: Placebo vs UMEC 250 µg QD; Test type: Superiority or Other; p = 0.683, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.5 to 2.3]
Statistical Analysis 6: Comparison: Placebo vs UMEC 15.6 µg BID; Test type: Superiority or Other; p = 0.456, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.2 to 2.7]
Statistical Analysis 7: Comparison: Placebo vs UMEC 31.25 µg BID; Test type: Superiority or Other; p = 0.399, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.7 to 1.1]

6. Primary Outcome: Change From Baseline in Diastolic Blood Pressure on Day 14 of Each Treatment Period
Description: Blood pressure measurement included diastolic blood pressure (DBP). Blood pressure was measured in a sitting position after the participant was kept at rest for at least 5 minutes. Analysis was performed using a mixed model, including treatment, period, period Baseline and mean Baseline for the measure as fixed effects and participant as a random effect. Baseline is the value recorded pre-dose on Day 1 of each treatment period; mean Baseline is the mean of the Baselines for each participant and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Change from Baseline was calculated as the assessment value at Day 14 minus the Baseline value.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 112 | 122 | 127 | 123 | 114 | 119 | 114 | 122
Millimeters of mercury (mmHg) | -2.1 (0.57) | -0.5 (0.55) | -0.8 (0.53) | -0.2 (0.54) | 0.3 (0.57) | 0.0 (0.55) | 0.6 (0.56) | -0.7 (0.55)
Statistical Analysis 1: Comparison: Placebo vs UMEC 15.6 µg QD; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [0.2 to 3.2]
Statistical Analysis 2: Comparison: Placebo vs UMEC 31.25 µg QD; Test type: Superiority or Other; p = 0.077, Mixed Models Analysis; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-0.1 to 2.8]
Statistical Analysis 3: Comparison: Placebo vs UMEC 62.5 µg QD; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [0.5 to 3.5]
Statistical Analysis 4: Comparison: Placebo vs UMEC 125 µg QD; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [0.9 to 3.9]
Statistical Analysis 5: Comparison: Placebo vs UMEC 250 µg QD; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [0.7 to 3.7]
Statistical Analysis 6: Comparison: Placebo vs UMEC 15.6 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [1.2 to 4.3]
Statistical Analysis 7: Comparison: Placebo vs UMEC 31.25 µg BID; Test type: Superiority or Other; p = 0.054, Mixed Models Analysis; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [0.0 to 3.0]

7. Primary Outcome: Change From Baseline in Pulse Rate on Day 14 of Each Treatment Period
Description: Pulse rate was measured in a sitting position after the participant was kept at rest for at least 5 minutes. Analysis was performed using a mixed model, including treatment, period, period Baseline and mean Baseline for the measure as fixed effects and participant as a random effect. Baseline is the value recorded pre-dose on Day 1 of each treatment period; mean Baseline is the mean of the Baselines for each participant and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Change from Baseline was calculated as the assessment value at Day 14 minus the Baseline value.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 112 | 122 | 127 | 123 | 114 | 119 | 114 | 122
Beats per minute | -0.4 (0.64) | -0.1 (0.62) | 1.2 (0.60) | 0.2 (0.61) | 0.2 (0.64) | 1.1 (0.62) | -0.4 (0.64) | -1.1 (0.62)
Statistical Analysis 1: Comparison: Placebo vs UMEC 15.6 µg QD; Test type: Superiority or Other; p = 0.752, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.4 to 2.0]
Statistical Analysis 2: Comparison: Placebo vs UMEC 31.25 µg QD; Test type: Superiority or Other; p = 0.072, Mixed Models Analysis; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.1 to 3.2]
Statistical Analysis 3: Comparison: Placebo vs UMEC 62.5 µg QD; Test type: Superiority or Other; p = 0.503, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.1 to 2.2]
Statistical Analysis 4: Comparison: Placebo vs UMEC 125 µg QD; Test type: Superiority or Other; p = 0.476, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.1 to 2.3]
Statistical Analysis 5: Comparison: Placebo vs UMEC 250 µg QD; Test type: Superiority or Other; p = 0.084, Mixed Models Analysis; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.2 to 3.2]
Statistical Analysis 6: Comparison: Placebo vs UMEC 15.6 µg BID; Test type: Superiority or Other; p = 0.970, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.8 to 1.7]
Statistical Analysis 7: Comparison: Placebo vs UMEC 31.25 µg BID; Test type: Superiority or Other; p = 0.423, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.4 to 1.0]

8. Primary Outcome: Change From Baseline in Albumin, Total Protein, and Hemoglobin on Day 14 of Each Treatment Period
Description: Blood samples were collected for the measurement of albumin, total protein, and hemoglobin at Baseline and Day 14. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70))
Population: ITT Population. Only those participants remaining in the study and contributing evaluable data for the indicated parameter were indicated by "n=X, X" in the category title and the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
Grams per liter (G/L)
  Albumin, n=111, 118, 120, 121, 112, 112, 112, 117 | -1.1 (2.46) | -1.0 (2.63) | -0.8 (2.47) | -0.9 (2.59) | -1.1 (2.65) | -1.0 (2.47) | -0.6 (2.41) | -0.7 (2.14)
  Total protein, n=111,118,120,121,112,112,112,117 | -1.9 (3.63) | -1.9 (3.83) | -1.4 (3.82) | -1.7 (3.48) | -1.9 (4.02) | -1.8 (3.58) | -1.1 (3.58) | -1.2 (3.09)
  Hemogloin, n=109,121,124,120,110,113,112,121 | -2.2 (7.24) | -2.8 (6.55) | -1.6 (6.66) | -2.3 (7.13) | -1.8 (7.44) | -1.4 (6.76) | -1.3 (6.59) | -2.0 (7.06)

9. Primary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Kinase (CK), Gamma Glutamyl Transferase (GGT) and Lactate Dehydrogenase (LDH) on Day 14 of Each Treatment Period
Description: Blood samples were collected for the measurement of ALP, ALT, AST, CK, GGT, and LDH at Baseline and Day 14. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: International Units/Liter (IU/L)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
International Units/Liter (IU/L)
  ALP, n=111, 118, 120, 121, 112, 112, 112, 117 | -0.7 (16.13) | -1.1 (14.35) | -1.8 (13.55) | -2.0 (10.73) | -2.8 (14.16) | -0.6 (10.90) | -0.6 (14.05) | -1.5 (9.88)
  ALT, n=111, 117, 120, 121, 112, 112, 112, 117 | 0.7 (12.15) | 0.6 (11.56) | 0.4 (11.24) | -0.1 (7.18) | -1.7 (8.44) | 1.4 (9.80) | 1.7 (16.17) | -1.3 (8.73)
  AST, n=110, 118, 120, 120, 112, 112, 112, 117 | 0.6 (7.53) | -0.3 (6.26) | 1.9 (18.69) | -0.4 (6.31) | -0.6 (7.51) | 0.7 (8.39) | 0.6 (7.24) | -0.3 (9.59)
  CK, n=111, 118, 120, 121, 112, 112, 112, 117 | 5.2 (69.94) | 6.3 (70.20) | 143.0 (1486.66) | -10.0 (73.53) | -2.5 (147.85) | 7.7 (105.96) | 6.9 (100.44) | 19.8 (284.94)
  GGT, n=111, 118, 120, 121, 112, 112, 112, 117 | 1.2 (15.06) | 0.7 (9.63) | 0.4 (10.63) | 0.0 (9.74) | -0.6 (8.31) | 0.2 (12.15) | 2.0 (10.18) | 0.9 (10.61)

10. Primary Outcome: Change From Baseline in Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, and Creatinine on Day 14 of Each Treatment Period
Description: Blood samples were collected for the measurement of direct bilirubin, indirect (ind) bilirubin, total bilirubin, and creatinine at Baseline and Day 14. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Micromoles/Liter (µM/L)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
Micromoles/Liter (µM/L)
  Direct bilirubin,n=111,118,120,121,112,112,112,117 | -0.2 (1.10) | -0.1 (1.10) | -0.1 (0.99) | -0.1 (0.95) | -0.1 (1.15) | -0.1 (1.15) | -0.1 (1.08) | -0.1 (1.10)
  Bilirubin, n=111,118,120,121,112,112,112,117 | -1.0 (3.94) | -0.9 (3.69) | -0.7 (3.36) | -0.9 (3.85) | -1.1 (5.15) | -0.9 (4.17) | -0.8 (4.19) | -0.9 (3.68)
  Ind Bilirubin, n=111,118,120,121,112,112,112,117 | -0.8 (3.42) | -0.8 (3.03) | -0.6 (2.93) | -0.8 (3.37) | -1.1 (4.42) | -0.8 (3.60) | -0.7 (3.63) | -0.8 (3.16)
  Creatinine, n=111,118,120,121,112,112,112,117 | 0.27 (9.218) | -0.67 (8.037) | -0.76 (6.242) | 0.94 (6.811) | -0.24 (7.450) | 0.15 (6.826) | 0.30 (7.297) | 0.22 (7.671)

11. Primary Outcome: Change From Baseline in Calcium, Chloride, Carbon Dioxide, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) on Day 14 of Each Treatment Period
Description: Blood samples were collected for the measurement of chloride, caron dioxide, glucose, potassium, sodium, and urea/BUN at Baseline and Day 14. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Micromoles/Liter (µM/L)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
Micromoles/Liter (µM/L)
  Chloride, n=111, 118, 120, 121, 112, 112, 112, 117 | 0.1 (2.11) | 0.4 (2.29) | 0.4 (2.29) | 0.3 (2.21) | 0.6 (2.18) | 0.3 (1.84) | 0.3 (2.22) | 0.3 (2.00)
  Carbon dioxide, n=110,118,120,120,112,112,112,117 | -0.6 (2.16) | -0.4 (2.73) | -0.6 (2.54) | -0.2 (2.88) | -0.4 (2.11) | -0.0 (2.55) | -0.5 (2.69) | -0.6 (2.38)
  Glucose, n=111, 118, 120, 121, 112, 112, 112, 117 | 0.01 (1.134) | 0.04 (0.975) | -0.15 (0.950) | 0.01 (1.012) | -0.29 (0.848) | -0.08 (1.048) | -0.09 (1.022) | -0.14 (0.778)
  Potassium, n=110, 118, 120, 120, 112, 112, 112,117 | 0.02 (0.400) | 0.05 (0.338) | 0.05 (0.416) | 0.03 (0.420) | 0.05 (0.353) | 0.02 (0.412) | 0.08 (0.387) | 0.09 (0.398)
  Sodium, n=111, 118, 120, 121, 112, 112, 112, 117 | -0.2 (1.78) | 0.2 (2.06) | -0.0 (2.14) | -0.2 (2.33) | -0.1 (1.99) | -0.3 (1.88) | -0.2 (2.23) | -0.4 (1.82)
  Urea/BUN, n=111, 118, 120, 121, 112, 112, 112, 117 | 0.11 (1.382) | 0.34 (1.149) | 0.02 (1.197) | 0.11 (1.283) | -0.04 (1.322) | 0.20 (1.303) | 0.02 (1.184) | 0.13 (1.265)

12. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils (ANC - Absolute Neutrophil Count), Platelet, and Leukocytes Count on Day 14 of Each Treatment Period
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, total neutrophils (ANC - Absolute neutrophil [neut] count), platelet, and leucocytes count at Day 14. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter (GI/L)
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
10^9 cells/Liter (GI/L)
  Basophil, n=109, 121, 124, 117, 110, 112, 111, 121 | 0.003 (0.0212) | -0.001 (0.0173) | -0.000 (0.0184) | 0.001 (0.0178) | 0.006 (0.0230) | -0.001 (0.0162) | -0.002 (0.0161) | 0.000 (0.0184)
  Eosinophils, n= 109, 121, 124, 117,110,112,111,121 | 0.097 (0.2400) | 0.023 (0.1988) | 0.029 (0.1928) | 0.036 (0.2056) | 0.036 (0.1944) | 0.039 (0.2583) | 0.040 (0.1799) | 0.039 (0.1862)
  Lymphocytes, n=109, 121, 124, 117,110,112,111,121 | -0.038 (0.5767) | -0.064 (0.5882) | -0.050 (0.5850) | -0.033 (0.4986) | -0.043 (0.5366) | -0.152 (0.5203) | -0.156 (0.5552) | -0.069 (0.6148)
  Monocytes, n=109, 121, 124, 117, 110, 112, 111,121 | 0.017 (0.1278) | 0.029 (0.1366) | 0.005 (0.1173) | 0.017 (0.1185) | 0.029 (0.1348) | 0.030 (0.1289) | 0.010 (0.1168) | -0.000 (0.1060)
  Total Neut, n= 109, 121, 124, 117, 110,112,111,121 | -0.204 (1.4615) | 0.032 (1.2279) | 0.119 (1.8710) | -0.175 (1.5228) | -0.161 (1.1780) | 0.107 (1.8329) | -0.133 (1.2785) | -0.080 (1.1597)
  Segmented Neut, n=109,121,124,117,110,112,111,121 | -0.204 (1.4615) | 0.032 (1.2279) | 0.119 (1.8710) | -0.175 (1.5228) | -0.161 (1.1780) | 0.107 (1.8329) | -0.133 (1.2785) | -0.080 (1.1597)
  Platelets,n=109, 121, 124, 119, 110, 112, 111, 119 | -1.4 (40.21) | -0.7 (30.35) | -1.0 (36.65) | -2.3 (36.32) | -2.1 (34.17) | -8.4 (40.89) | -2.2 (33.07) | -1.0 (39.34)
  Leukocytes,n=109,121,124, 117, 110, 112, 111, 121 | -0.12 (1.740) | 0.01 (1.385) | 0.10 (1.867) | -0.15 (1.664) | -0.14 (1.400) | 0.02 (1.913) | -0.24 (1.423) | -0.11 (1.402)

13. Primary Outcome: Change From Baseline in the Percentage of Basophils, Eosinophils, Lymphocytes, Monocytes, and Segmented Neutrophils in Blood on Day 14 of Each Treatment Period
Description: Blood samples were collected for the measurement of the percentage of basophils, eosinophils, lymphocytes, monocytes, and segmented neutrophils (neut) at Baseline and Day 14. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of cells in blood
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
Percentage of cells in blood
  Basophils, n=109,121,124,117,111,112,111,121 | 0.05 (0.302) | -0.01 (0.240) | -0.02 (0.273) | 0.03 (0.286) | 0.08 (0.318) | 0.00 (0.212) | -0.02 (0.248) | 0.00 (0.268)
  Eosinophils, n= 109,121,124,117,110,112,111,121 | 1.45 (3.380) | 0.30 (2.782) | 0.32 (2.896) | 0.68 (3.100) | 0.56 (2.403) | 0.55 (3.142) | 0.65 (2.537) | 0.56 (2.481)
  Lymphocytes, n=109,121,124,117,110,112,111,121 | -0.00 (6.861) | -0.64 (7.590) | -0.29 (7.485) | 0.62 (8.069) | -0.06 (6.996) | -1.97 (8.203) | -0.76 (8.001) | -0.46 (7.650)
  Monocytes, n=109,121,124,117,110,112,111,121 | 0.30 (1.735) | 0.45 (1.941) | 0.04 (1.798) | 0.41 (1.787) | 0.52 (1.719) | 0.45 (1.622) | 0.43 (2.626) | 0.07 (1.585)
  Neutrophils, n=109,121,124,117,110,112,111,121 | -1.80 (8.264) | -0.11 (8.872) | -0.04 (8.739) | -1.73 (9.048) | -1.11 (8.107) | 0.96 (9.319) | -0.30 (9.252) | -0.17 (8.676)
  Segmented Neut, n=109,121,124,117,110,112,111,121 | -1.80 (8.264) | -0.11 (8.872) | -0.04 (8.739) | -1.73 (9.048) | -1.11 (8.107) | 0.96 (9.319) | -0.30 (9.252) | -0.17 (8.676)

14. Primary Outcome: Change From Baseline in Hematocrit on Day 14 of Each Treatment Period
Description: Blood samples were collected for the measurement of hematocrit (proportion of red blood cells in blood) at Baseline and Day 14. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 109 | 121 | 124 | 120 | 110 | 113 | 112 | 121
Proportion of red blood cells in blood | -0.0093 (0.02298) | -0.0118 (0.02180) | -0.0075 (0.02271) | -0.0092 (0.02198) | -0.0082 (0.02452) | -0.0079 (0.02053) | -0.0084 (0.02259) | -0.0087 (0.02279)

15. Primary Outcome: Number of Participants for the Indicated Urinalysis Parameters Tested by Dipstick on Day 14 of Each Treatment Period
Description: Urinalysis parameters included: Urine Bilirubin (UB), Urine Occult Blood (UOB), Urine Glucose (UG), Urine Ketones (UK), Urine Nitrite (UN), Urine Protein (UP), and Urine Leukocyte Esterase test for detecting White Blood Cell (UWBC). The dipstick was a strip used to detect the presence or absence of these parameters in the urine sample. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative (Neg), Trace (T), 1+, 2+, and 3+, and for UG the result can be read as Neg, T, T or 1/10 G/dL, 1+ or 1/4 G/dL, 3+ or 1 G/dL, indicating proportional concentrations in the urine sample. Data are reported as the number of participants who had neg, T, 1+, 2+ and 3+ levels at Day 14.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70))
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
Participants
  UB, Neg, n=109,121,125,120,112, 113,112,119 | 109 | 121 | 125 | 120 | 112 | 112 | 112 | 119
  UOB, T, n=109,121,125,120,112,113,112,119 | 8 | 8 | 14 | 12 | 13 | 11 | 8 | 13
  UOB, 1+, n=109,121,125,120,112,113,112,119 | 5 | 8 | 4 | 5 | 5 | 7 | 5 | 2
  UOB, 2+, n=109,121,125,120,112,113,112,119 | 5 | 1 | 3 | 2 | 0 | 1 | 3 | 2
  UOB, 3+, n=109,121,125,120,112,113,112,119 | 6 | 3 | 1 | 1 | 4 | 3 | 2 | 3
  UOB, Neg, n=109,121,125,120,112,113,112,119 | 85 | 101 | 103 | 100 | 90 | 91 | 94 | 99
  UG, T, n=109,121,125,120,112,113,112,119 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
  UG, T or 1/10, n=109,121,125,120,112,113,112,119 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  UG, 1+ or 1/4, n=109,121,125,120,112,113,112,119 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  UG, 3+ or 1, n=109,121,125,120,112,113,112,119 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  UG, Neg, n=109,121,125,120,112,113,112,119 | 107 | 118 | 124 | 119 | 112 | 112 | 111 | 119
  UK, T, n=109,121,125,120,112,113,112,119 | 4 | 3 | 5 | 2 | 8 | 0 | 2 | 3
  UK, Neg, n=109,121,125,120,112,113,112,119 | 103 | 118 | 119 | 116 | 104 | 112 | 110 | 113
  UK, 1+, n=109,121,125,120,112,113,112,119 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  UK, 2+, n=109,121,125,120,112,113,112,119 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  UK, 3+, n=109,121,125,120,112,113,112,119 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  UN, Neg, n=109,121,125,120,112,113,112,119 | 97 | 113 | 116 | 108 | 108 | 109 | 103 | 105
  UN, Pos, n=109,121,125,120,112,113,112,119 | 12 | 8 | 9 | 12 | 4 | 4 | 9 | 14
  UP, Neg, n=109,121,125,120,112,113,112,119 | 99 | 112 | 110 | 116 | 102 | 108 | 107 | 111
  UP, T, n=109,121,125,120,112,113,112,119 | 4 | 6 | 8 | 2 | 6 | 3 | 4 | 4
  UP, 1+, n=109,121,125,120,112,113,112,119 | 4 | 2 | 6 | 1 | 4 | 2 | 1 | 4
  UP, 2+, n=109,121,125,120,112,113,112,119 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  UWBC, Neg, n=109,121,125,120,112,113,112,119 | 88 | 96 | 100 | 90 | 82 | 88 | 89 | 85
  UWBC, T, n=109,121,125,120,112,113,112,119 | 6 | 5 | 6 | 11 | 8 | 5 | 5 | 11
  UWBC, 1+, n=109,121,125,120,112,113,112,119 | 6 | 9 | 12 | 12 | 12 | 12 | 4 | 10
  UWBC, 2+, n=109,121,125,120,112,113,112,119 | 4 | 8 | 5 | 3 | 5 | 8 | 11 | 12
  UWBC, 3+, n=109,121,125,120,112,113,112,119 | 5 | 3 | 2 | 3 | 5 | 0 | 3 | 1

16. Primary Outcome: Urine pH on Day 14 of Each Treatment Period
Description: Urine samples were collected for the measurement of urine pH by dipstick method at Day 14. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0).
Time Frame: Day 14 of each treatment period (up to Study Day 70)
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 109 | 121 | 125 | 120 | 112 | 113 | 112 | 119
Scores on a scale | 5.89 (0.635) | 5.97 (0.709) | 6.05 (0.718) | 6.07 (0.743) | 5.90 (0.678) | 5.99 (0.720) | 5.89 (0.690) | 5.90 (0.684)

17. Primary Outcome: Urine Specific Gravity on Day 14 of Each Treatment Period
Description: Urine samples were collected for the measurement of urine specific gravity by dipstick method at Day 14. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. A urinary specific gravity measurement is a routine part of urinalysis. The reference range is 1.002-1.030.
Time Frame: Day 14 of each treatment period (up to Study Day 70)
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 109 | 121 | 125 | 120 | 112 | 113 | 112 | 118
Ratio | 1.0194 (0.00703) | 1.0198 (0.00628) | 1.0194 (0.00732) | 1.0185 (0.00653) | 1.0201 (0.00780) | 1.0192 (0.00707) | 1.0189 (0.00734) | 1.0193 (0.00671)

18. Primary Outcome: Number of Participants With the Indicated Abnormal Electrocardiogram Findings
Description: Electrocardiograph measurements performed at Screening (Visit 1) and at Day 1 and Day 14 (pre-dose, 10 minutes post-dose and 2 hours post-dose.of each treatment period). Any clinically significant findings were identified during participant monitoring.
Time Frame: Day 14 of each treatment period (up to Study Day 70)
Population: ITT Population. Only those participants remaining in the study and contributing evaluable data at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
Participants
  Conduction | 14 | 17 | 10 | 12 | 10 | 11 | 7 | 12
  Depolarisation/Repolarisation(QRS-T) | 21 | 20 | 26 | 20 | 32 | 25 | 22 | 28
  Myocardial Infarction | 2 | 3 | 1 | 2 | 1 | 0 | 1 | 2
  P-Wave and QRS Morphology | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
  Rhythm | 12 | 13 | 15 | 12 | 13 | 15 | 17 | 21

19. Primary Outcome: Number of Participants With the Indicated 24 Hour Holter Findings
Description: Twenty-four hour Holter ECG measurements were obtained using a 12-lead Holter monitor. The Holter monitor is worn by the participant for 24 hours, and the monitor continuously records the heart's rhythm while the monitor is worn. Following the 24-hour period, the data from the monitor were downloaded and transmitted to the centralized vendor for analysis and interpretation by a licensed cardiologist. The 24-hour Holter ECG measurements were obtained at during the screening period and on Day 14 of each treatment period. The number of participants with clinically significant change (abnormal or normal) were reported.
Time Frame: Day 14 of each treatment period (up to Study Day 70)
Population: ITT Population. Only participants with sufficient data (at least 16 hours of recorded data) at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 41 | 41 | 51 | 46 | 46 | 42 | 39 | 49
Participants
  Abnormal | 6 | 3 | 7 | 7 | 8 | 8 | 7 | 7
  Normal | 35 | 38 | 44 | 39 | 38 | 34 | 32 | 42

20. Secondary Outcome: Change From Baseline (BL) in the Weighted Mean (WM) 0-24 Hour FEV1 Obtained Post-AM Dose on Day 14 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The WM FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. Baseline is the 0h value obtained prior to the AM dose on Day 14 of the treatment period. Change from BL at a was calculated as WM at the evaluated time point minus BL. Analysis was performed using a mixed model, including treatment, period, period Baseline FEV1, and mean Baseline FEV1 as fixed effects and participant as a random effect.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 33 | 35 | 49 | 42 | 45 | 38 | 35 | 43
Liters | -0.025 (0.0255) | 0.060 (0.0249) | 0.077 (0.0222) | 0.092 (0.0232) | 0.094 (0.0229) | 0.048 (0.0243) | 0.097 (0.0252) | 0.043 (0.0231)

21. Secondary Outcome: Change in Baseline in Serial FEV1 Over 0-24 Hours After the Morning Dose on Day 14 of Each Treatment Period
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Serial FEV1 measurements were taken electronically by spirometry. Serial FEV1 was measured at 5, 15, 30 minutes (min), 1, 3, 6, 9, 12, 16, 20, 23 and 24 hours (h) post-dose. Baseline is the 0h value obtained prior to the AM dose on Day 14 of the treatment period. Change from Baseline was calculated as FEV1 value at the evaluated time point minus Baseline. Analysis was preformed using a repeated measures model with terms for period, treatment, time, mean Baseline, period Baseline, and time by mean Baseline, time by period Baseline, and time by treatment interactions.
Time Frame: Baseline and Day 14 of each treatment period (up to Study Day 70)
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
Liters
  5 min, n=41, 39, 49, 46, 44, 42, 38, 48 | 0.024 (0.0329) | 0.095 (0.0330) | 0.110 (0.0296) | 0.077 (0.0309) | 0.123 (0.0312) | 0.042 (0.0326) | 0.141 (0.0338) | 0.118 (0.0301)
  15 min, n=41, 41, 51, 46, 46, 42, 39, 49 | 0.002 (0.0322) | 0.082 (0.0322) | 0.124 (0.0290) | 0.090 (0.0303) | 0.115 (0.0305) | 0.038 (0.0320) | 0.160 (0.0331) | 0.108 (0.0294)
  30 min, n=45, 42, 39, 49, 45, 42, 39, 49 | 0.012 (0.0318) | 0.109 (0.0317) | 0.115 (0.0285) | 0.092 (0.0299) | 0.149 (0.0301) | 0.040 (0.0315) | 0.158 (0.0326) | 0.110 (0.0290)
  1 h, n=41, 41, 51, 46, 46, 42, 39, 49 | 0.025 (0.0319) | 0.127 (0.0318) | 0.161 (0.0286) | 0.143 (0.0300) | 0.165 (0.0302) | 0.113 (0.0316) | 0.164 (0.0327) | 0.168 (0.0291)
  3 h, n=41, 41, 51, 46, 46, 42, 39, 49 | 0.000 (0.0353) | 0.141 (0.0353) | 0.175 (0.0317) | 0.156 (0.0332) | 0.143 (0.0335) | 0.143 (0.0350) | 0.182 (0.0362) | 0.165 (0.0322)
  6 h, n=41, 40, 51, 46, 46, 42, 39, 48 | 0.007 (0.0368) | 0.099 (0.0369) | 0.089 (0.0330) | 0.108 (0.0346) | 0.134 (0.0349) | 0.076 (0.0365) | 0.157 (0.0378) | 0.100 (0.0337)
  9 h, n=41, 40, 51, 46, 46, 42, 39, 49 | -0.049 (0.0354) | 0.043 (0.0356) | 0.061 (0.0318) | 0.118 (0.0333) | 0.117 (0.0335) | 0.081 (0.0351) | 0.072 (0.0363) | 0.075 (0.0323)
  12 h, n=41, 41, 51, 46, 46, 41, 39, 49 | -0.044 (0.0395) | 0.015 (0.0394) | 0.021 (0.0354) | 0.060 (0.0372) | 0.056 (0.0374) | 0.016 (0.0393) | 0.050 (0.0405) | 0.056 (0.0360)
  16 h, n=40, 40, 51, 46, 46, 42, 38, 49 | -0.074 (0.0408) | 0.006 (0.0407) | 0.022 (0.0364) | 0.052 (0.0382) | 0.035 (0.0384) | 0.008 (0.0402) | 0.053 (0.0419) | 0.009 (0.0370)
  20 h, n=40, 41, 51, 45, 46, 41, 39, 49 | -0.149 (0.0441) | -0.046 (0.0438) | -0.003 (0.0393) | 0.057 (0.0415) | 0.029 (0.0416) | -0.050 (0.0437) | -0.005 (0.0450) | -0.012 (0.0400)
  23 h, n=40, 40, 51, 46, 46, 42, 39, 48 | 0.013 (0.0391) | 0.033 (0.0390) | 0.056 (0.0349) | 0.107 (0.0366) | 0.087 (0.0369) | 0.058 (0.0386) | 0.081 (0.0399) | 0.037 (0.0356)
  24 h, n=41, 41, 51, 45, 46, 42, 39, 49 | 0.039 (0.0387) | 0.105 (0.0386) | 0.110 (0.0347) | 0.143 (0.0366) | 0.139 (0.0366) | 0.088 (0.0384) | 0.187 (0.0397) | 0.124 (0.0353)

22. Secondary Outcome: Change From Baseline in Mean Morning (AM) and Evening (PM) Pre-treatment Peak Expiratory Flow (PEF) Over Day 7 to Day 14 of Each Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants daily in the morning and evening just prior to each dose, using an electronic peak flow meter, throughout the 14-day Treatment Period. Only the averaged daily AM and PM PEF over Days 7 to 14 was analyzed. The analysis was performed using a mixed effects analysis of covariance model with fixed effect terms for treatment and period; Baseline PEF AM and PM, gender and age fitted as covariates; and participant as a random effect.
Time Frame: Baseline (Day 7 prior to each treatment period) and the last 7 days of each treatment period (up to Study Day 70)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 126 | 131 | 138 | 133 | 128 | 135 | 126 | 133
Liters per minute
  AM, n=112, 120, 125, 122, 113, 116, 110, 122 | 0.8 (31.98) | 5.2 (42.17) | 1.7 (37.95) | 1.1 (31.23) | 6.4 (32.31) | 6.4 (43.24) | 5.0 (35.82) | 5.8 (33.00)
  PM, n=116, 123, 123, 119, 115, 118, 108, 121 | -5.1 (34.43) | 10.0 (43.47) | 1.5 (37.95) | -0.9 (31.32) | 9.8 (31.25) | 9.3 (40.03) | 2.5 (35.89) | 8.7 (30.55)

23. Secondary Outcome: Change From Baseline in the Mean Number of Puffs Per Day of Rescue Albuterol/Salbutamol Over Day 7 to Day 14 of Each Treatment Period
Description: The mean number of puffs per day of rescue salbutamol at Baseline (i.e. run-in or washout data) and on-treatment were recorded. Total puffs was calculated as (Number of Puffs + (2 x number of Nebules)). Only the 7 days proceeding each treatment period were included in the Baseline calculations. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 7 prior to each treatment period) and the last 7 days of each treatment period (up to Study Day 70)
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Number of puffs
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.25 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Number analyzed (Participants) | 109 | 117 | 119 | 114 | 108 | 111 | 105 | 118
Number of puffs | -0.3 (1.25) | -0.4 (1.42) | -0.2 (1.06) | -0.3 (1.14) | -0.4 (1.19) | -0.3 (1.31) | -0.6 (1.49) | -0.3 (1.04)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the end of treatment (up to Study Day 70).
Description: On-treatment SAEs and non-serious AEs were collected in members of the ITT Population, comprised of all participants who had received at least one dose of randomized study medication during treatment period. Provision was made for the collection of any SAEs during the 9 - 14 days screening (pre-treatment) period. None was reported.
Groups:
- UMEC 31.5 µg QD: Participants received UMEC 31.25 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
Arm/Group | Placebo | UMEC 15.6 µg QD | UMEC 31.5 µg QD | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 15.6 µg BID | UMEC 31.25 µg BID
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/131 | 0/138 | 0/133 | 0/128 | 1/135 | 0/126 | 0/133
Other Adverse Events (participants affected / at risk) | 4/126 | 7/131 | 7/138 | 12/133 | 11/128 | 12/135 | 7/126 | 7/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=126) | UMEC 15.6 µg QD (N=131) | UMEC 31.5 µg QD (N=138) | UMEC 62.5 µg QD (N=133) | UMEC 125 µg QD (N=128) | UMEC 250 µg QD (N=135) | UMEC 15.6 µg BID (N=126) | UMEC 31.25 µg BID (N=133)
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=126) | UMEC 15.6 µg QD (N=131) | UMEC 31.5 µg QD (N=138) | UMEC 62.5 µg QD (N=133) | UMEC 125 µg QD (N=128) | UMEC 250 µg QD (N=135) | UMEC 15.6 µg BID (N=126) | UMEC 31.25 µg BID (N=133)
Headache (Nervous system disorders) | 2 | 5 | 4 | 5 | 4 | 6 | 2 | 6
Nasopharyngitis (Infections and infestations) | 1 | 3 | 0 | 1 | 3 | 1 | 4 | 2
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 5 | 0 | 1 | 1 | 0
Product taste abnormal (General disorders) | 0 | 0 | 2 | 1 | 4 | 5 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.